CLINICAL TRIAL: NCT04411459
Title: Risk Factors for Prolonged Invasive Mechanical Ventilation in COVID-19 Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Azienda Usl di Bologna (Other Government)
Collaborators: Lorenzo Gamberini (Unknown)
Responsible Party: Sponsor
Other Study IDs: 273/2020/OSS/AUSLBO
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: COVID-19; Mechanical Ventilation; Quality of Life; Radiologic Increased Density of Lung; Sedation; Complication of Treatment
Keywords: COVID-19; Mechanical Ventilation; Quality of life; Complications during ICU stay
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 pneumonia patients: Patients needing intubation and mechanical ventilation for COVID-19 related pneumonia without other primary causes of ICU admission
  Interventions: Other: Invasive mechanical ventilation

INTERVENTIONS:
Other: Invasive mechanical ventilation — Invasive mechanical ventilation for respiratory failure associated to COVID-19 pneumonia

SUMMARY:
This multicentric prospective clinical practice study aims at evaluating clinical factors associated with a prolonged invasive mechanical ventilation and other outcomes such as mortality and ICU length of stay in patients affected from COVID-19 related pneumonia and ARDS.

DETAILED DESCRIPTION:
Background

On February 21th 2020, SARS-CoV-2 outbreak erupted in Italy and, in the immediately subsequent period, all the Italian regional Health Systems had to face with an overwhelming increase of COVID-19 admissions requiring isolation, oxygen, ventilation and ICU beds.

The COVID-19 related pneumonia presented as a particular entity in terms of clinical management and different ICUs adopt different clinical strategies, sometimes this is due to the local resources' availability. Mortality rate of the patients admitted to ICU is up to 26%.

To date, it is not clear which clinical, pharmacological and radiologic factors relate to a prolonged duration of mechanical ventilation, mortality and ICU length of stay and it's urgent to understand these aspects in order to develop optimal strategies to allow faster but safe paths for these patients.

Hypothesis and significance

SARS-CoV-2 related pneumonia ICU management is still undefined, in fact this entity seems to have clinical aspects rather different from other forms of interstitial pulmonary syndromes evolving in diffuse alveolar damage and many aspects related to ventilation such pulmonary compliance, driving pressure and response to pronation are very different from what traditionally observed from other forms of ARDS, moreover an abnormal trend towards hypercoagulability has been described in these patients.

Different treatments have been proposed and are under evaluation such as Tocilizumab, corticosteroids, hydroxychloroquine, antivirals, anticoagulants and antiplatelet therapies.

These treatments, together with common ICU practice aspects such as early/late tracheostomy, ventilatory parameters believed adequate in order to start a weaning procedure, fluidic balance, choice of analgesia and sedation regimens, are not standardized in this particular syndrome due to the lack of evidence available and there is need for information about which factors correlate to a lower duration of mechanical ventilation and mortality.

Collected data:

* Demographics and anamnesis: age, sex, weight, height, previous pathologies (Hypertension, Chronic ischemic heart disease, Chronic kidney disease, COPD, Diabetes, Chronic liver disease, active cancer, immunosuppressive therapy), smoker status, therapy with ACE-inhibitors, statins and Angiotensin II Receptor Blockers.
* Conditions at ICU admission: date of symptoms onset (fever and or cough), date of hospital admission, date of ICU admission, SOFA and SAPS II score, high flow nasal oxygen therapy before intubation, NIV/CPAP trial before intubation, duration of the NIV/CPAP trial, PaO2/FiO2 value before intubation, initial tidal volume set, initial PEEP set, Initial pplateau observed.
* Ventilation during the first 5 days: lowest PaO2/FiO2 value, ventilatory strategy (pressure control ventilation vs volume control ventilation and volumes), lowest static respiratory system compliance, highest driving pressure, highest PEEP, highest arterial pCO2 observed, number and duration of pronation cycles, response in terms of oxygenation to the first pronation, need for decapneization, use of nitric oxide, tracheostomy date, need for extracorporeal membrane oxygenation treatment.
* Pharmacologic strategies during the first 5 days: sedative regimen and maximum doses, neuromuscular blocking agents (type of NMBA and duration of continuous infusion).
* COVID specific therapies: antivirals (type, start and end date), chloroquine, tocilizumab (start date and route of administration), intravenous corticosteroids, other specific therapies.
* Other supportive therapies: first line antibacterial regimen, amines (maximum dose), renal replacement therapy, fluidic balance during the first 3 days after ICU admission, anticoagulation, antiaggregation.
* Complications during ICU stay:

  * Cardiovascular (myocardial infarction, new onset supraventricular or ventricular arrhythmia, pulmonary embolism, pulmonary edema, haemorragic shock, cardiogenic shock, acute peripheral ischemia, pneumothorax)
  * Neurologic (new onset ischemic stroke or cerebral haemorrage, critical illness polyneuropathy / myopathy, new onset seizures)
  * Gastroenteric (gastrointestinal bleeding, severe diarrhea, intestinal occlusion, gastrointestinal perforation/ischemia)
  * Extrapulmonary infections (documented blood steam, urinary tract, central nervous system, abdominal infection)
  * Pulmonary infections after intubation (early onset VAP - < 7 days of mechanical ventilation, late onset VAP - ≥ 7 days of mechanical ventilation)
* Weaning from mechanical ventilation: last day of highest PEEP, first attempt of pressure support ventilation (PSV), P/F at the first attempt of PSV, entity of pressure support at the first attempt of PSV, PEEP at the first attempt of PSV, day of extubation, non-invasive ventilation or high flow oxygen therapy after extubation, first day of spontaneous breathing, need for reintubation and date
* Radiology: first available CT, last CT before ICU admission and intubation, last ICU follow-up CT. First available chest X ray, last chest X ray before ICU admission and intubation, last ICU- follow up chest X ray. 30 days follow-up CT (if available).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ICU admission because of the need of mechanical ventilation in the context of COVID-19 related pneumonia (swab proven)

Exclusion Criteria:

* COVID-19 related pneumonia complicating the clinical course of patients admitted to the ICU for another reason (e.g. trauma, stroke)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolls patients admitted to ICU needing intubation and mechanical ventilation bacause of respiratory failure for COVID-19 pneumonia without other primary causes for ICU admission
Sampling Method: Non-Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Duration of mechanical ventilation and 28 days ventilator free days | 28 days
  Ventilator free days (VFDs) will be calculated in a time frame of 28 days, the beginning of observation will coincide with the day of intubation and observation will end after successful disconnection from mechanical ventilation.
  For intubated patients, post extubation non invasive ventilation (NIV) will not be accounted as a ventilation period, in case of interval reintubation within 28 days, VFDs will be counted from the last successful extubation.
  For tracheostomized patients, ventilator free days will be counted after successful disconnection from mechanical ventilation and interval reconnections will be considered in the ventilation interval as for intubated patients.

SECONDARY OUTCOMES:
ICU Mortality | 60 days
30 days survival after ICU discharge | 30 days
90 days survival after ICU discharge | 90 days
Quality of life at 90 days after ICU discharge measured with 15D instrument | 90 days
  15D instrument (http://www.15d-instrument.net/15d/) will be administered via telephonic interview
  Areas assessed: MOBILITY, VISION, HEARING, BREATHING, SLEEPING, EATING, SPEECH, EXCRETION, USUAL ACTIVITIES, MENTAL FUNCTION, DISCOMFORT AND SYMPTOMS, DEPRESSION, DISTRESS, VITALITY, SEXUAL ACTIVITY
Radiologic aspects - structured description of CT and RX data | 90 days
  First available CT, last CT before ICU admission and intubation, last ICU follow-up CT. First available chest X ray, last chest X ray before ICU admission and intubation, last ICU- follow up chest X ray and 30 days follow-up CT (if available) will be evaluated, if available.
  Structured description
  CT scan
  Date: yyyy/mm/dd Parenchymal alterations: ground glass, crazy paving, parenchymal consolidation Extension: monolateral, bilateral Number of lobes involved: (1-5) Percentage of parenchymal involvement: 0-100% Distribution: subpleural, random, diffuse
  X-ray scan
  Date: yyyy/mm/dd Main aspects: normal, focal lesions, monolateral multifocal lesions (right/left), diffuse multifocal lesions Lesion aspects: interstitial, interstitial/alveolar, alveolar, consolidations Pleural effusion presence and entity
  Pulmonary involvement score:
  0 = no involvement
  1. =< 25%
  2. = 25-50% 3= 50-75%
  4 => 75% Total score (0-6): score of the right lung + score of the left lung
Quality of life at 1 year after ICU discharge and persistent symptoms | 1 year
  15D instrument (http://www.15d-instrument.net/15d/) will be administered via telephonic interview
  Areas assessed: MOBILITY, VISION, HEARING, BREATHING, SLEEPING, EATING, SPEECH, EXCRETION, USUAL ACTIVITIES, MENTAL FUNCTION, DISCOMFORT AND SYMPTOMS, DEPRESSION, DISTRESS, VITALITY, SEXUAL ACTIVITY
  Persistent symptoms explored: Dyspnea measured with mMRC scale, palpitations, cough, arthromyalgia
Radiologic aspects at 1 year CT scan | 1 year
  Presence and extension of pulmonary fibrosing and non fibrosing signs
Pulmonary function tests at 1 year - FEV1% | 1 year
  FEV1% - Forced expiratory volume 1 second, % of predicted value referred to normative population
Pulmonary function tests at 1 year - FVC% | 1 year
  FVC% - Forced vital capacity, % of predicted value referred to normative population
Pulmonary function tests at 1 year - FEV1/FVC% | 1 year
  FEV1/FVC% - Forced expiratory volume 1 second/Forced Vital capacity, % of predicted value referred to normative population
Pulmonary function tests at 1 year - | 1 year
  DLCO% - Diffusing capacity for carbon monoxide, % of predicted value referred to normative population

CONTACTS AND LOCATIONS:
Locations (20):
- Italy (20):
  - Ospedale Santa Maria Annunziata - Anestesia e Rianimazione, Bagno a Ripoli, FI
  - A.O. SS. Antonio, Biagio e Cesare Arrigo - Anestesia e Rianimazione, Alessandria
  - Anestesia e Rianimazione - Ospedale Civile di Baggiovara, Baggiovara
  - Anestesia e Rianimazione - Ospedale di Bentivoglio, Bentivoglio
  - Azienda Unità Sanitaria Locale, Bologna
  - Anestesia e Rianimazione - Ospedale Bellaria, Bologna
  - Anestesia e Rianimazione - Policlinico Universitario S.Orsola - Malpighi, Bologna
  - Anestesia e Terapia intensiva dei trapianti addominali e chirurgia epatobiliare - Policlinico Universitario S.Orsola - Malpighi, Bologna
  - Anestesia e Terapia Intensiva Polivalente - Policlinico Universitario S.Orsola - Malpighi, Bologna
  - Ospedale SS. Trinità - Anestesia e Rianimazione, Borgomanero
  - Anestesia e Rianimazione - Ospedale M. Bufalini, Cesena
  - Anestesia e Rianimazione - Ospedale degli Infermi, Faenza
  - Anestesia e Rianimazione Universitaria - Arcispedale Sant'Anna Ferrara, Ferrara
  - Anestesia e Rianimazione - Ospedale Morgagni - Pierantoni, Forlì
  - Anestesia e Rianimazione - Ospedale di Imola S.Maria della Scaletta, Imola
  - Ospedale Santo Stefano - Anestesia e Rianimazione, Prato
  - Anestesia e Rianimazione - Ospedale S. Maria delle Croci, Ravenna
  - Anestesia e Rianimazione - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Anestesia e Rianimazione - Ospedale di Riccione, Riccione
  - Anestesia e Rianimazione - Ospedale Infermi, Rimini

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yehya N, Harhay MO, Curley MAQ, Schoenfeld DA, Reeder RW. Reappraisal of Ventilator-Free Days in Critical Care Research. Am J Respir Crit Care Med. 2019 Oct 1;200(7):828-836. doi: 10.1164/rccm.201810-2050CP. PMID 31034248
- [Background] Gattinoni L, Chiumello D, Caironi P, Busana M, Romitti F, Brazzi L, Camporota L. COVID-19 pneumonia: different respiratory treatments for different phenotypes? Intensive Care Med. 2020 Jun;46(6):1099-1102. doi: 10.1007/s00134-020-06033-2. Epub 2020 Apr 14. No abstract available. PMID 32291463
- [Result] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Result] Bhatraju PK, Ghassemieh BJ, Nichols M, Kim R, Jerome KR, Nalla AK, Greninger AL, Pipavath S, Wurfel MM, Evans L, Kritek PA, West TE, Luks A, Gerbino A, Dale CR, Goldman JD, O'Mahony S, Mikacenic C. Covid-19 in Critically Ill Patients in the Seattle Region - Case Series. N Engl J Med. 2020 May 21;382(21):2012-2022. doi: 10.1056/NEJMoa2004500. Epub 2020 Mar 30. PMID 32227758
- [Result] Richardson S, Hirsch JS, Narasimhan M, Crawford JM, McGinn T, Davidson KW; the Northwell COVID-19 Research Consortium; Barnaby DP, Becker LB, Chelico JD, Cohen SL, Cookingham J, Coppa K, Diefenbach MA, Dominello AJ, Duer-Hefele J, Falzon L, Gitlin J, Hajizadeh N, Harvin TG, Hirschwerk DA, Kim EJ, Kozel ZM, Marrast LM, Mogavero JN, Osorio GA, Qiu M, Zanos TP. Presenting Characteristics, Comorbidities, and Outcomes Among 5700 Patients Hospitalized With COVID-19 in the New York City Area. JAMA. 2020 May 26;323(20):2052-2059. doi: 10.1001/jama.2020.6775. PMID 32320003
- [Derived] Dalpiaz G, Gamberini L, Carnevale A, Spadaro S, Mazzoli CA, Piciucchi S, Allegri D, Capozzi C, Neziri E, Bartolucci M, Muratore F, Coppola F, Poerio A, Giampalma E, Baldini L, Tonetti T, Cappellini I, Colombo D, Zani G, Mellini L, Agnoletti V, Damiani F, Gordini G, Laici C, Gola G, Potalivo A, Montomoli J, Ranieri VM, Russo E, Taddei S, Volta CA, Scaramuzzo G. Clinical implications of microvascular CT scan signs in COVID-19 patients requiring invasive mechanical ventilation. Radiol Med. 2022 Feb;127(2):162-173. doi: 10.1007/s11547-021-01444-7. Epub 2022 Jan 16. PMID 35034320
- [Derived] Gamberini L, Mazzoli CA, Prediletto I, Sintonen H, Scaramuzzo G, Allegri D, Colombo D, Tonetti T, Zani G, Capozzi C, Dalpiaz G, Agnoletti V, Cappellini I, Melegari G, Damiani F, Fusari M, Gordini G, Laici C, Lanza MC, Leo M, Marudi A, Papa R, Potalivo A, Montomoli J, Taddei S, Mazzolini M, Ferravante AF, Nicali R, Ranieri VM, Russo E, Volta CA, Spadaro S; ICU-RER COVID-19 Collaboration; Radiology Collaborators (to be indexed and searchable into PubMed); Pneumology Collaborators (to be indexed and searchable into PubMed). Health-related quality of life profiles, trajectories, persistent symptoms and pulmonary function one year after ICU discharge in invasively ventilated COVID-19 patients, a prospective follow-up study. Respir Med. 2021 Nov-Dec;189:106665. doi: 10.1016/j.rmed.2021.106665. Epub 2021 Oct 22. PMID 34717097
- [Derived] Gamberini L, Mazzoli CA, Sintonen H, Colombo D, Scaramuzzo G, Allegri D, Tonetti T, Zani G, Capozzi C, Giampalma E, Agnoletti V, Becherucci F, Bertellini E, Castelli A, Cappellini I, Cavalli I, Crimaldi F, Damiani F, Fusari M, Gordini G, Laici C, Lanza MC, Leo M, Marudi A, Nardi G, Ottaviani I, Papa R, Potalivo A, Ranieri VM, Russo E, Taddei S, Volta CA, Spadaro S; ICU-RER COVID-19 Collaboration. Quality of life of COVID-19 critically ill survivors after ICU discharge: 90 days follow-up. Qual Life Res. 2021 Oct;30(10):2805-2817. doi: 10.1007/s11136-021-02865-7. Epub 2021 May 12. PMID 33977415
- [Derived] Gamberini L, Tonetti T, Spadaro S, Zani G, Mazzoli CA, Capozzi C, Giampalma E, Bacchi Reggiani ML, Bertellini E, Castelli A, Cavalli I, Colombo D, Crimaldi F, Damiani F, Fogagnolo A, Fusari M, Gamberini E, Gordini G, Laici C, Lanza MC, Leo M, Marudi A, Nardi G, Ottaviani I, Papa R, Potalivo A, Russo E, Taddei S, Volta CA, Ranieri VM; ICU-RER COVID-19 Collaboration. Factors influencing liberation from mechanical ventilation in coronavirus disease 2019: multicenter observational study in fifteen Italian ICUs. J Intensive Care. 2020 Oct 15;8:80. doi: 10.1186/s40560-020-00499-4. eCollection 2020. PMID 33078076